CLINICAL TRIAL: NCT00655408
Title: Iron-Deficiency Anemia in Infants: Comparative Study of Two Weekly Supplement Programs
Brief Title: Iron-Deficiency Anemia in Infants in Two Weekly Programs
Acronym: IDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sao Jose do Rio Preto Medical School (Other)
Responsible Party: Sao Jose do Rio Preto Medical School, Sao Jose do Rio Preto Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAMERP-001
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2008-04-09 (Estimated); Status verified 2008-04

CONDITIONS: Anemia
Keywords: Infants; Prevalence; Iron; Deficiency; Treatment
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator): For infants with ages between six and 24 months, iron supplementation is the main treatment for iron deficiency.This study was carried out using two intervention groups. All children received 12 weekly doses of 25 mg of elemental iron.
  Group 1 administered in the government healthcare clinic. Group 2 administered children's home.
  The study showed treatment compliance in both groups.
  Interventions: Drug: elemental iron

INTERVENTIONS:
Drug: elemental iron — Iron supplementation.
  Other Names: doses of 25 mg of elemental iron

SUMMARY:
This work aims at establishing the effectiveness of weekly doses of ferrous sulfate administered by mothers compared with weekly supplements administered directly by healthcare professionals, to reducing anemia prevalence.

DETAILED DESCRIPTION:
Some studies have shown satisfactory results in reducing the prevalence of iron deficiency using weekly doses of ferrous sulfate, thereby avoiding these side effects. This deficiency is the most common nutritional disorder during childhood and does not only affect individuals from developing countries but also those from industrialized nations.

For infants with ages between six and 24 months, iron supplementation is the main treatment for iron deficiency. In this age range the prevalence of anemia is at least 20%. However, studies have shown a low rate of compliance by mothers during the recommended period, which may be caused by a lack of care or, more probably, due to the side effects caused by long-term daily ferrous sulfate supplementation, which include nausea, vomiting, diarrhea, staining of teeth and abdominal pain.

This specific study is randomized clinical trial study, achieved in a government healthcare clinic in Sao Jose do Rio Preto, Sao Paulo, Brazil. This study was carried out using two intervention groups. All children received 12 weekly doses of 25 mg of elemental iron, either administered in the government healthcare clinic or at the children's home.

The study showed treatment compliance in both groups. Prevalence of anemia for all children was 75% at the beginning of supplementation and 46.3% at the end of the period (p < 0.0005). Reduction rate for anemic children was 38.3%. Average increases in hemoglobin concentration levels were 0.75 g/dL and 0.65 g/dL, respectively, for home interventions and healthcare clinic administration (p < 0.00005).

ELIGIBILITY:
Inclusion Criteria:

* Ages ranging between six and 24 months old

Exclusion Criteria:

* Positive results for the Guthrie test
* Use of ferrous sulfate supplements
* Infections process at the time of first consultation

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2003-04; Primary Completion 2003-09 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Test (serum hemoglobin) | assessed at the before of the treatment period

SECONDARY OUTCOMES:
Test (serum hemoglobin) | assessed after 12 weekly with iron supplement

CONTACTS AND LOCATIONS:
Overall Officials: Coutinho Geraldo Gaspar Paes Leme, MD, Principal Investigator — University Medical School f São Jose do Rio Preto-Brazil

REFERENCES:
- [Derived] Coutinho GG, Goloni-Bertollo EM, Pavarino-Bertelli EC. Effectiveness of two programs of intermittent ferrous supplementation for treating iron-deficiency anemia in infants: randomized clinical trial. Sao Paulo Med J. 2008 Nov;126(6):314-8. doi: 10.1590/s1516-31802008000600004. PMID 19274317